CLINICAL TRIAL: NCT03916224
Title: Clinical Practice and Risk Factors for Major Adverse Events in the Tracheal Intubation in the Intensive Care Unit: A Prospective Multicentre Study
Brief Title: Adverse Events in the Tracheal Intubation in the Intensive Care Unit
Acronym: INTUPROS
Status: Completed | Type: Observational
Sponsor: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 1149-N-18
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2019-04

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication; Intubation
Keywords: Intubation; Airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intubated critically ill patients: Critically ill patients older than 18 years old, intubated in an Intensive Care Unit.

SUMMARY:
The airway management is essential in the Critical Care setting, both normal and difficult airway patients. Intubation is a risk procedure in which a great number of complications may occur, including death. The poor physiological reserve of critical patients may suppose an additional handicap to carry out successfully intubation.

The purpose of this study is to analyze the prevalence and risk factors for major complications in the intubation process in the Intensive Care Unit (ICU). In addition, the investigators will assess the impact of preoxygenation and the use of videolaryngoscope on the occurrence of major and minor complications. Finally, this study will review the drug protocols used in each participant ICU during intubation process.

DETAILED DESCRIPTION:
The correct airway and difficult airway management are essential in the Critical Care setting.

Intubation is a procedure frequently carried out by intensivist and a great number of complications have been related. Serious complications can occur, including the development of severe hypoxemia, arrhythmias, cardiac arrest with permanent anoxic brain damage or death. Additionally the poor physiological reserve of critically ill patients and the variable operator experience, means that this technique must be considered a risk event in critical patients.

In recent years, it has been taken more and more importance of preoxygenation as a strategy that can avoid major complications in the intubation process.

Similarly, the use of devices that facilitate intubation such as videolaryngoscopy, has been included in difficult airway management protocols. If the use of videolaryngoscopy compared with traditional laryngoscopy is associated with a higher success rate and a lower incidence of complications, still remains controversial.

The investigators want to know the prevalence and risk factors for major complications in the intubation process of patients admitted to Intensive Care Unit (ICU). In addition, this study will try to assess the use and impact of both preoxygenation and videolaryngoscope in the intubation process.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are intubated at the participating Intensive Care Units.

Exclusion Criteria:

* Intubations carried out at other different areas.
* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients, older than 18 years old, that are intubated at the participating Units.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of major complications in the intubation process of patients admitted to Intensive Care Units. | 28 days
  This study will analyze the prevalence of major complications related to intubation technique in the participant critical care units. This information will be useful in order to determinate the risk factors associated.

SECONDARY OUTCOMES:
Number of minor complications in the intubation process of patients admitted to Intensive Care Units. | 28 days
  This study will analyze the prevalence of minor complications related to intubation technique in the participant critical care units. This information will be useful in order to determinate the risk factors associated.
Number of episodes in which pre-oxygenation methods are used | 28 days
  Pre-oxygenation is considered a strategy that can avoid complications in the intubation process. The investigators will define the frequency of use in each participant unit and its association with the development of major and minor complications. The study will describe the different pre-oxygenation options: conventional ambu mask, non invasive ventilation, high flow oxygenation.
Frequency of videolaryngoscope use to perform intubation technique. | 28 days
  Nowadays the videolaryngoscopy is an useful tool included in difficult airway management protocols. Despite of this, the benefit associated to the videolaryngoscopy employment compared with traditional laryngoscopy is controversial.
  The investigators will analyze its role in the intubation protocols and the factors that determine its use. The difficult airway predictors scales used in the participant units are: Cormack-Lehane, MACOCHA.
Association between videolaryngoscope use and incidence of complications compared with conventional laryngoscopy. | 28 days
  Nowadays, the videolaryngoscopy is an useful tool included in difficult airway management protocols. Despite of this, the benefit associated to the videolaryngoscopy employment compared with traditional laryngoscopy is controversial.
  The investigator will analyze (adjusting for confounding variables) if the use of videolaryngoscope is associated with a lower incidence of major and minor complications compared with conventional laryngoscopy.
Occurrence of major complications in the intubation process of patients admitted to Intensive Care Units comparing COVID and non-COVID patients 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose Garnacho-Montero, MD,Phd, Principal Investigator — Virgen Macarena University Hospital
Locations (1):
- Jose Garnacho-Montero, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Scheduled teleconferences
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From now to the end of analysis
Access Criteria: All participants